CLINICAL TRIAL: NCT02872922
Title: Effects of Therapeutic Ultrasound on Endothelial Function of Patients With Type 2 Diabetes Mellitus: Randomized Clinical Trial
Brief Title: Effects of Low Intensity Therapeutic Ultrasound on Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Luis Ulisses Signori, PhD, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UFSM1
Record Dates: First submitted 2016-08-11; First posted 2016-08-19 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Endothelial function; Ultrasonic Therapy; Vascular endothelium; Nitric oxide; Ultrasound
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ultrasonic Therapy; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Endothelial function after CWUT (Active Comparator): Endothelial function of the all patients before and after application continuous waveform of ultrasound therapy (CWUT) measured by technique flow-mediated dilation (FMD).
  Interventions: Other: Low intensity therapeutic ultrasound
- Endothelial function after PWUT (Active Comparator): Endothelial function of the all patients before and after application pulsed waveform of ultrasound therapy (PWUT) measured by technique flow-mediated dilation (FMD).
  Interventions: Other: Low intensity therapeutic ultrasound
- Endothelial function after PLACEBO (Active Comparator): In the placebo intervention, all of the procedures above are repeated, but with the ultrasound equipment powered off. Endothelial function of the all patients before and after application placebo waveform of ultrasound therapy measured by technique flow-mediated dilation (FMD)
  Interventions: Other: Low intensity therapeutic ultrasound

INTERVENTIONS:
Other: Low intensity therapeutic ultrasound — The ultrasound equipment (Sonopulse III, 1 MHz, IBRAMED, Brazil) was calibrated with the radiation force method. In study, the head of the transducer will be positioned and applied for 5 min over the brachial artery at the same point that will be evaluated the endothelium function (Cruz et al., 2016). Continuous waveforms of ultrasound therapy (CWUT) are applied in the stationary mode for 5 minutes at a spatial averaged temporal intensity (SATA) of 0.4 W/cm2 using a transducer 1-MHz. A pulsed waveform of ultrasound therapy (PWUT) are applied (5 minutes) with a 20% duty cycle (2 ms on, 8 ms off), which represents a constant intensity of 0.08 W/cm2 SATA. In the placebo intervention, all of the procedures above are repeated, but with the ultrasound equipment powered off (Cruz et al., 2016).
  Other Names: Ultrasonic therapy, Ultrasound

SUMMARY:
Endothelium is a cell layer that interposes blood and smooth muscle of vessels. This biological sensor reacts to physical and chemical stimuli by synthesis and/or liberation of regulatory substances like nitric oxide (NO), which acts on vascular tone, growth of muscle cells and platelet aggregation and leukocyte. Clinically, endothelial function measured by technique flow-mediated dilation (FMD) is a strong predictor of cardiovascular events and all-cause mortality. Previo study demonstrated that continuous and pulsed therapeutic 1-MHz ultrasound waveforms improved endothelial function in health volunteers and this vasodilation persisted for 20 min, which provided them with anti-inflammatory vascular effects. In subjects with type 2 diabetes (DM2) the chronical hyperglycemia and dyslipidemia reduce NO bioavailability causing endothelial dysfunction. Low intensity therapeutic ultrasound is an electrotherapeutic instrument employed in musculoskeletal injuries that promotes endothelium-dependent vasodilation, and its mechanism of action has not been studied on DM2. The aim of our study is evaluate endothelial function of patients with DM2 after different waveforms (placebo, continuous and pulsed) of therapeutic ultrasound. Therapeutic ultrasound is a electrotherapeutic instrument that can changes arterial endothelial function of subjects with DM2 because of NO bioavailability increasing, which implies anti-inflammatory and vasodilatory beneficial alterations for diabetic patients.

DETAILED DESCRIPTION:
Evaluation of endothelial function will be made by flow-mediated dilation (FMD). The therapeutic ultrasound will applied over brachial artery using continuous (CUT: 0,4W/cm2), pulsed (PUT: 20% duty cycle, 0,08W/cm2SATA) and Placebo (equipment off) waveforms during 5min in 3 intercalated days.

ELIGIBILITY:
Inclusion Criteria:

* The subjects that joined the study will be alphabetized volunteers
* Age between 25 and 65 years old,
* Absence of morbid obesity,
* Non-smokers,
* With no symptoms of skeletal muscle disorders,
* No previous performing cardiovascular surgery,
* No previous diagnose of rheumatic, neurological, oncological, immune or hematologic diseases,
* Without evidence of psychiatric diseases and/or cognitive deficit.

Exclusion Criteria:

* Insulin dependent diabetes
* Leukocytosis, impaired fasting glycemia (<70 and >300 mg/dL) and
* Brachial artery diameter less than 2.5mm and larger than 5.0mm.
* On the day of the assessments have consumed of the alcoholic drink, caffeine and citrus juice

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-12-10 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Percentage of the endothelium-dependent vasodilation (%FMD) | Five minutes after application of therapeutic ultrasound
  Vessel diameter responses to reactive hyperemia are expressed as percentage change in relation to diameter before cuff inflation (%FMD = [(hyperemia maximum diameter - baseline precuff diameter)/(baseline precuff diameter)] / 100) (Corretti et al. 2002; Thijssen et al. 2011).
  Baseline precuff diameter is expressed in millimeter (mm). Hyperemia maximum diameter is expressed in millimeter (mm). Arterial endothelium-dependent vasodilation are evaluated by technique flow-mediated dilation (FMD) with high-resolution vascular ultrasound and a 5- to 12-MHz linear transducer (Logiq P6, GE Healthcare, GE Ultrasound Korea), according to the American Heart Association Guidelines (Corretti et al. 2002), with adjustments (Thijssen et al. 2011).

SECONDARY OUTCOMES:
Percentage of the endothelium-independent vasodilation (%NMD) | Five minutes after application of therapeutic ultrasound
  Endothelium-independent vasodilation is measured after sublingual nitroglycerin (NMD) spray (0.4 mg). Vessel diameter responses nitroglycerin are expressed as percentage change in relation to diameter before cuff inflation and before drug administration (%NMD = [(nitroglycerin maximum diameter - baseline precuff diameter)/(baseline precuff diameter)] / 100) (Corretti et al. 2002; Iida et al. 2006; Thijssen et al. 2011). Baseline precuff diameter is expressed in millimeter (mm) and Nitroglycerin maximum diameter is expressed in millimeter (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Luis U Signori, PhD, Principal Investigator — Universidade Federal de Santa Maria
Locations (1):
- Universidade Federal do Rio Grande, Rio Grande, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Poredos P, Jezovnik MK. Testing endothelial function and its clinical relevance. J Atheroscler Thromb. 2013;20(1):1-8. doi: 10.5551/jat.14340. Epub 2012 Sep 10. PMID 22972428
- [Background] Shechter M, Shechter A, Koren-Morag N, Feinberg MS, Hiersch L. Usefulness of brachial artery flow-mediated dilation to predict long-term cardiovascular events in subjects without heart disease. Am J Cardiol. 2014 Jan 1;113(1):162-7. doi: 10.1016/j.amjcard.2013.08.051. Epub 2013 Oct 5. PMID 24169007
- [Background] Thijssen DH, Black MA, Pyke KE, Padilla J, Atkinson G, Harris RA, Parker B, Widlansky ME, Tschakovsky ME, Green DJ. Assessment of flow-mediated dilation in humans: a methodological and physiological guideline. Am J Physiol Heart Circ Physiol. 2011 Jan;300(1):H2-12. doi: 10.1152/ajpheart.00471.2010. Epub 2010 Oct 15. PMID 20952670
- [Background] Xu Y, Arora RC, Hiebert BM, Lerner B, Szwajcer A, McDonald K, Rigatto C, Komenda P, Sood MM, Tangri N. Non-invasive endothelial function testing and the risk of adverse outcomes: a systematic review and meta-analysis. Eur Heart J Cardiovasc Imaging. 2014 Jul;15(7):736-46. doi: 10.1093/ehjci/jet256. Epub 2014 Jan 7. PMID 24399339
- [Result] Cruz JM, Hauck M, Cardoso Pereira AP, Moraes MB, Martins CN, da Silva Paulitsch F, Plentz RD, Peres W, Vargas da Silva AM, Signori LU. Effects of Different Therapeutic Ultrasound Waveforms on Endothelial Function in Healthy Volunteers: A Randomized Clinical Trial. Ultrasound Med Biol. 2016 Feb;42(2):471-80. doi: 10.1016/j.ultrasmedbio.2015.10.002. Epub 2015 Nov 12. PMID 26578361